CLINICAL TRIAL: NCT01069705
Title: A Phase III Open-Label Extension Study to Assess the Safety and Efficacy of Tobramycin Inhalation Powder After Manufacturing Process Modifications (TIPnew) in Cystic Fibrosis (CF) Patients Who Successfully Completed Participation in Study CTBM100C2303E1
Brief Title: Second Open Label Extension to Bridging Study CTBM100C2303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100C2303E2
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Infections; Pseudomonas Aeruginosa
Keywords: Tobramycin Inhalation Powder; Cystic fibrosis; Lung diseases; Anti-Bacterial Agents; Treatment of pulmonary infections with P. aeruginosa in cystic fibrosis participants
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tobramycin Inhalation Powder (TIPnew) (Experimental): Participants received four capsules of 28 mg TIPnew (112 mg), inhaled twice a day (b.i.d.) in the morning and the evening given in a cycle of 28 days on treatment followed by 28 days off treatment for three consecutive cycles.
  Interventions: Drug: Tobramycin inhalation powder

INTERVENTIONS:
Drug: Tobramycin inhalation powder — Tobramycin dry powder for inhalation in capsules administered by the T-326 inhaler.

SUMMARY:
This was an open-label, single arm (uncontrolled) study in participants suffering from cystic fibrosis, who have completed their study participation in CTBM100C2303 and extension study one CTBM100C2303E1 (all visits), who were proven infected with Pseudomonas aeruginosa at enrollment into CTBM100C2303.

ELIGIBILITY:
Inclusion Criteria:

* Completed all visits in study CTBM100C2303 and CTBM100C2303E1, and visit 11 of study CTBM100C2303E1 took place not more than 5 days before enrollment into this study.
* Confirmed diagnosis of cystic fibrosis participants with P. aeruginosa infection.
* Forced Expiratory Volume in one second (FEV1) at screening (at start of study CTBM100C2303) must be between 25% and 80% of normal predicted values.

Exclusion Criteria:

* Any use of inhaled anti-pseudomonal antibiotics between the termination of the trial CTMB100C2303E1 and the enrollment into this study.
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02-12 (Actual); Primary Completion 2012-03-19 (Actual); Study Completion 2012-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Riga, Latvia
- Lithuania (2):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Durban, South Africa

REFERENCES:
- [Result] Konstan MW, Flume PA, Galeva I, Wan R, Debonnett LM, Maykut RJ, Angyalosi G. One-year safety and efficacy of tobramycin powder for inhalation in patients with cystic fibrosis. Pediatr Pulmonol. 2016 Apr;51(4):372-8. doi: 10.1002/ppul.23358. Epub 2015 Dec 27. PMID 26709158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centres in 8 countries from 12 February 2010 to 19 March 2012.
Pre-assignment Details: This study enrolled 49 Participants with Cystic Fibrosis who completed participation in the study CTBM100C2303E1 (NCT00982930).
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Started | 49
Completed | 46
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who completed their participation in C2303E1, who gave their consent to enter the extension 2 study and who received at least one dose of study drug in the extension 2 study.
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug.
Time Frame: From time of first administration of study drug until study completion (up to 169 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
Participants | 23

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: From time of consent to 4 weeks after study completion (up to 199 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
Participants | 2

3. Primary Outcome: Percentage of Participants With a Decrease of ≥20% in Forced Expiratory Value in One Second (FEV1) Percent (%) Predicted From Pre-dose to 30-minute Post-dose
Description: Airway Reactivity >= 20% relative decrease in FEV1% predicted from pre-dose to 30 minutes post-dose. Relative Change = 100 * (30 minutes Post-dose - Pre-dose)/Pre-dose assessed by the number and percentage of participants with a decrease of ≥ 20% in FEV1 % predicted from pre-dose to 30 minutes post-dose.
Time Frame: Pre-dose and post-dose of Day 1 and Day 29 of every Cycle (5, 6, 7)
Population: Safety population included all participants who completed their participation in C2303E1, who gave their consent to enter the extension 2 study and who received at least one dose of study drug in the extension 2 study. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
percentage of participants
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 5 (Day 1): number analyzed (Participants) | 44
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 5 (Day 1) | 2.3
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 5 (Day 29): number analyzed (Participants) | 45
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 5 (Day 29) | 0.0
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 6 (Day 1): number analyzed (Participants) | 40
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 6 (Day 1) | 2.5
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 6 (Day 29): number analyzed (Participants) | 46
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 6 (Day 29) | 4.3
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 7 (Day 1): number analyzed (Participants) | 45
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 7 (Day 1) | 6.7
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 7 (Day 29): number analyzed (Participants) | 45
  Acute Change from Pre-dose to 30 mins Post-dose Cycle 7 (Day 29) | 0.0

4. Primary Outcome: Percentage of Participants With Frequency Decrease From Baseline in the Post-baseline Audiology Tests
Description: Auditory acuity of participants was measured using a standard dual-channel audiometer at frequencies from 250 to 8000 Hertz, and an audiogram (pure-tone air conduction) and tympanogram were performed by an audiologist. The categories reported includes >= 10dB decrease in 3 consecutive frequencies in either ear, >= 15dB decrease in 2 consecutive frequencies in either ear, and >= 20dB decrease in at least one frequency in either ear
Time Frame: Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: All participants included in the safety population with at least one audiology testing. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 19
percentage of participants
  Cycle 5: Day 1; >= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 13
  Cycle 5: Day 1; >= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 0.0
  Cycle 5: Day 1; >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 13
  Cycle 5: Day 1; >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear | 0.0
  Cycle 5: Day 1; >= 20 dB Decrease in at least one Frequency in Either Ear: number analyzed (Participants) | 13
  Cycle 5: Day 1; >= 20 dB Decrease in at least one Frequency in Either Ear | 0.0
  Cycle 5: Day 29; >= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 0.0
  Cycle 5: Day 29; >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear | 5.3
  Cycle 5: Day 29; >= 20 dB Decrease in at least one Frequency in Either Ear | 0.0
  Cycle 6: Day 29; >= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 0.0
  Cycle 6: Day 29; >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear | 5.3
  Cycle 6: Day 29; >= 20 dB Decrease in at least one Frequency in Either Ear | 0.0
  Cycle 7: Day 29; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 10.5
  Cycle 7: Day 29; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 5.3
  Cycle 7: Day 29; >= 20 dB Decrease in at Least One Frequency in Either Ear | 5.3
  Follow Up: Week 57/Day 57; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 5
  Follow Up: Week 57/Day 57; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 20.0
  Follow Up: Week 57/Day 57; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 5
  Follow Up: Week 57/Day 57; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 0.0
  Follow Up: Week 57/Day 57; >= 20 dB Decrease in at Least One Frequency in Either Ear: number analyzed (Participants) | 5
  Follow Up: Week 57/Day 57; >= 20 dB Decrease in at Least One Frequency in Either Ear | 0.0

5. Secondary Outcome: Relative Change From Baseline of Forced Expiratory Volume in One Second (FEV1) Percent Predicted to Each Post-baseline Visit
Description: Forced expiratory volume in one second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 % predicted was a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. Relative change in FEV1 % predicted from baseline to pre-dose day X = ((pre-dose day X FEV1 % predicted - baseline FEV1 % predicted) / baseline FEV1 % predicted) x 100.
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in FEV1 % predicted
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
percent change in FEV1 % predicted
  Baseline: number analyzed (Participants) | 48
  Baseline | 59.5 (16.51)
  Relative Change from Baseline to Cycle 5 (Day 1): number analyzed (Participants) | 46
  Relative Change from Baseline to Cycle 5 (Day 1) | 11.4 (21.79)
  Relative Change from Baseline to Cycle 5 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 5 (Day 29) | 12.6 (24.49)
  Relative Change from Baseline to Cycle 6 (Day 1): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 6 (Day 1) | 8.6 (19.73)
  Relative Change from Baseline to Cycle 6 (Day 29): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 6 (Day 29) | 11.9 (24.23)
  Relative Change from Baseline to Cycle 7 (Day 1): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 7 (Day 1) | 9.0 (22.44)
  Relative Change from Baseline to Cycle 7 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 7 (Day 29) | 10.1 (26.37)
  Relative Change from Baseline to Follow -Up (Week 57/Day 57): number analyzed (Participants) | 42
  Relative Change from Baseline to Follow -Up (Week 57/Day 57) | 8.1 (25.79)

6. Secondary Outcome: Relative Change From Baseline of Forced Vital Capacity (FVC) Percent Predicted to Each Post-baseline Visit
Description: Percent Predicted Forced Vital Capacity (FVC%) is the maximal exhaled breath volume following a maximal inhaled breath. Overall change in percent predicted FVC = (observed value)/(predicted value) * 100%. A higher value indicates a greater response.
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in FVC % predicted
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
percent change in FVC % predicted
  Baseline: number analyzed (Participants) | 48
  Baseline | 75.0 (17.63)
  Relative Change from Baseline to Cycle 5 (Day 1): number analyzed (Participants) | 46
  Relative Change from Baseline to Cycle 5 (Day 1) | 5.1 (15.60)
  Relative Change from Baseline to Cycle 5 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 5 (Day 29) | 5.2 (17.87)
  Relative Change from Baseline to Cycle 6 (Day 1): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 6 (Day 1) | 2.6 (16.36)
  Relative Change from Baseline to Cycle 6 (Day 29): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 6 (Day 29) | 6.2 (20.01)
  Relative Change from Baseline to Cycle 7 (Day 1): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 7 (Day 1) | 2.3 (19.20)
  Relative Change from Baseline to Cycle 7 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 7 (Day 29) | 2.9 (20.40)
  Relative Change from Baseline to Follow-up (Week 57/Day 57): number analyzed (Participants) | 42
  Relative Change from Baseline to Follow-up (Week 57/Day 57) | 4.0 (20.37)

7. Secondary Outcome: Relative Change From Baseline of Forced Expiratory Flow Rate Over 25 and 75 Percent (FEF25-75%) Predicted to Each Post-baseline Visit
Description: Forced Expiratory Flow Rate Over 25 and 75 Percent (FEF25-75%) is the forced expiratory flow from 25% to 75% of the Forced Vital Capacity (FVC). Relative change in FEF25-75% from baseline to pre-dose day X = (pre-dose day X FEF25-75 - baseline FEF25-75) / baseline FEF25-75) • 100.
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in (FEF25-75)% predicted
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
percent change in (FEF25-75)% predicted
  Baseline: number analyzed (Participants) | 48
  Baseline | 36.8 (20.30)
  Relative Change from Baseline to Cycle 5 (Day 1): number analyzed (Participants) | 46
  Relative Change from Baseline to Cycle 5 (Day 1) | 37.7 (57.39)
  Relative Change from Baseline to Cycle 5 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 5 (Day 29) | 43.2 (67.51)
  Relative Change from Baseline to Cycle 6 (Day 1): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 6 (Day 1) | 35.1 (66.39)
  Relative Change from Baseline to Cycle 6 (Day 29): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 6 (Day 29) | 34.3 (63.53)
  Relative Change from Baseline to Cycle 7 (Day 1): number analyzed (Participants) | 45
  Relative Change from Baseline to Cycle 7 (Day 1) | 44.4 (80.91)
  Relative Change from Baseline to Cycle 7 (Day 29): number analyzed (Participants) | 44
  Relative Change from Baseline to Cycle 7 (Day 29) | 36.1 (61.75)
  Relative Change from Baseline to Follow-up (Week 57/Day 57): number analyzed (Participants) | 42
  Relative Change from Baseline to Follow-up (Week 57/Day 57) | 35.6 (77.34)

8. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Sputum Density to Each Post-baseline Visit
Description: Pseudomonas Aeruginosa Density refers to overall density, defined as the sum of Biotypes (mucoid, dry and small colony variant). Absolute change was determined using the formula; Change = Post-baseline value- baseline value. Absolute Change in Pseudomonas Aeruginosa Sputum density is measured in log 10 Colony Forming Units per gram (Log 10 CFU/g).
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10 CFU/g
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
Log 10 CFU/g
  Baseline: number analyzed (Participants) | 45
  Baseline | 7.4 (1.50)
  Change from Baseline to Cycle 5 (Day 1): number analyzed (Participants) | 37
  Change from Baseline to Cycle 5 (Day 1) | -1.1 (2.82)
  Change from Baseline to Cycle 5 (Day 29): number analyzed (Participants) | 40
  Change from Baseline to Cycle 5 (Day 29) | -3.7 (2.95)
  Change from Baseline to Cycle 6 (Day 1): number analyzed (Participants) | 41
  Change from Baseline to Cycle 6 (Day 1) | -1.6 (2.95)
  Change from Baseline to Cycle 6 (Day 29): number analyzed (Participants) | 41
  Change from Baseline to Cycle 6 (Day 29) | -3.6 (2.73)
  Change from Baseline to Cycle 7 (Day 1): number analyzed (Participants) | 39
  Change from Baseline to Cycle 7 (Day 1) | -1.5 (3.40)
  Change from Baseline to Cycle 7 (Day 29): number analyzed (Participants) | 40
  Change from Baseline to Cycle 7 (Day 29) | -2.6 (2.92)
  Change from Baseline to Follow-up (Week 57/Day 57): number analyzed (Participants) | 18
  Change from Baseline to Follow-up (Week 57/Day 57) | -1.8 (3.62)

9. Secondary Outcome: Change From Baseline in Tobramycin Minimum Inhibitory Concentration (MIC) Values for Pseudomonas Aeruginosa to Each Post-baseline Visit
Description: Minimum Inhibitory Concentration (MIC) is defined as the lowest concentration of an antimicrobial agent required to inhibit the visible growth of a microorganism after overnight incubation.
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29) and Follow-up (Week 57/Day 57)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram/millilitre
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
microgram/millilitre
  Baseline | 2.2 (9.11)
  Change from Baseline in Cycle 5 (Day 1): number analyzed (Participants) | 36
  Change from Baseline in Cycle 5 (Day 1) | 31.4 (117.6)
  Change from Baseline in Cycle 5 (Day 29): number analyzed (Participants) | 30
  Change from Baseline in Cycle 5 (Day 29) | 21.6 (92.35)
  Change from Baseline in Cycle 6 (Day 1): number analyzed (Participants) | 39
  Change from Baseline in Cycle 6 (Day 1) | 39.3 (138.37)
  Change from Baseline in Cycle 6 (Day 29): number analyzed (Participants) | 35
  Change from Baseline in Cycle 6 (Day 29) | 25.5 (94.74)
  Change from Baseline in Cycle 7 (Day 1): number analyzed (Participants) | 36
  Change from Baseline in Cycle 7 (Day 1) | 3.7 (22.94)
  Change from Baseline in Cycle 7 (Day 29): number analyzed (Participants) | 38
  Change from Baseline in Cycle 7 (Day 29) | 31.7 (115.97)
  Change from Baseline to Follow-up (Week 57/Day 57): number analyzed (Participants) | 19
  Change from Baseline to Follow-up (Week 57/Day 57) | 1.7 (11.14)

10. Secondary Outcome: Number of Participants Who Used New Antipseudomonal Antibiotic During Treatment Period
Description: The rate of anti-pseudomonal antibiotics use were determined from the collection of concomitant medication during the study Treatment period.
Time Frame: Baseline, Cycles 5, 6, 7 (Days 1, 29)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
Participants | 7

11. Secondary Outcome: Percentage of Participants With Hospitalization Due to Respiratory Serious Adverse Events (SAEs)
Description: as for outcome 2
Time Frame: From time of consent to 4 weeks after study completion (up to 199 days)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
percentage of participants | 4.1

12. Secondary Outcome: Number of Days of Hospitalization Due to Respiratory Serious Adverse Events (SAEs)
Description: The average number of days patients were hospitalized due to respiratory events during the study.
Time Frame: From time of consent to 4 weeks after study completion (up to 199 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
Number analyzed (Participants) | 49
days | 16.5 (2.12)

ADVERSE EVENTS:
Time Frame: From the time of first administration of study drug until study completion (up to 169 days)
Description: AEs were deemed treatment-emergent if the onset date was on or after the date of the first study drug of extension 2 and until study completion of the extension 2.
Arm/Group | Tobramycin Inhalation Powder (TIPnew)
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 2/49
Other Adverse Events (participants affected / at risk) | 22/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIPnew) (N=49)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIPnew) (N=49)
Hypoacusis (Ear and labyrinth disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 1
Acute sinusitis (Infections and infestations) | 2
Alcaligenes infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Burkholderia cepacia complex infection (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 5
Respiratory tract infection viral (Infections and infestations) | 4
Antibiotic resistant Staphylococcus test positive (Investigations) | 1
Protein urine present (Investigations) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.